CLINICAL TRIAL: NCT01196130
Title: Assessment of Targeted Therapy Against Colorectal Cancer (ATTACC) Screening Protocol
Brief Title: Colorectal Cancer Umbrella Protocol - Assessment of Targeted Therapies Against Colorectal Cancer (ATTACC Program) Screening Protocol
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2009-0091; R01CA172670 (NIH); RP110584 (Other Grant/Funding Number: CPRIT); NCI-2017-00505 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
Keywords: Metastatic colorectal cancer; CRC; Colorectal adenocarcinoma; Biomarker determination; Tumor tissue; Treatment protocols
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (16 mL) collected and archived tumor samples (primary tumor or metastatic site) from prior surgeries or biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biomarker Assessment: Leftover sample of tumor tissue from a previous procedure used for biomarker testing. Blood drawn for biomarker testing, to check for levels of cytokines, and to check the circulating tumor cells (CTCs). Cancer Symptom Questionnaire completion about cancer symptoms.
  Interventions: Behavioral: Cancer Symptom Questionnaire; Other: Biomarker Testing

INTERVENTIONS:
Behavioral: Cancer Symptom Questionnaire — 5 minute questionnaire(s) completed at each study visit.
Other: Biomarker Testing — Blood draw at each study visit for biomarker and cytokine testing.

SUMMARY:
The goal of this clinical research study is to test for biomarkers in patients with metastatic or unresectable, locally advanced colorectal cancer. Biomarkers are chemical "markers" in the tumor tissue and/or blood that may be related to your reaction to cancer drugs.

This is an investigational study. This study's biomarker testing is for research purposes only.

Up to 1280 patients will be enrolled in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
The effectiveness of drugs used to treat colorectal cancer may be different from person to person. Researchers want to learn if certain biomarkers can be used to help predict which cancer drugs may work better than other drugs in different people with colorectal cancer.

Study Participation:

If you agree to take part in this study, the following tests and procedures will be performed:

* A leftover sample of tumor tissue from a previous procedure, if available, will be used for biomarker testing.
* Blood (about 3 tablespoons) will be drawn for biomarker testing, to check for levels of cytokines (proteins that may affect the immune system), and to check the circulating tumor cells (CTCs) in your blood.
* You will be asked how well you are able to perform the normal activities of daily living (performance status).

You will also fill out a questionnaire about the cancer symptoms. This should take about 5 minutes.

Biomarker Test Results:

The study doctor and staff will review the biomarker test results with you.

If the results seem to show that a certain investigational drug may help to control the cancer, and the drug is available through a separate MD Anderson clinical research study called a "companion" drug study, your doctor may recommend that you have additional tests and procedures performed. The tests and procedures will be performed as part of the companion drug study to see if you are eligible to receive that drug. You will be asked to sign a separate consent form for the companion drug study.

It is possible that the biomarker test results may seem to show that more than one drug may help to control the cancer. If so, it may be possible that you could receive the other drug(s) under other companion studies in the future. The study tests described below would be repeated during those other studies as well.

Even if the biomarker testing shows that a certain drug may be helpful, it is possible that you may not be eligible to take part in the separate companion drug study, the study drug may not be available, or there may be other reasons you cannot take part in the drug study. You may also decide that you do not want to take part in the companion drug study. Your doctor will discuss other available treatment options with you.

Study Visits:

At study visits for this biomarker research study, the following tests and procedures will be performed:

* You will fill out the cancer symptom questionnaire.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for biomarker, cytokine, and CTC testing.

Your schedule of study visits will depend on whether or not you take part in a companion study. There is a different schedule of visits for participants who do not take part in a companion study but instead either take part in a clinical research study that is not a companion study or they receive standard cancer drug(s).

If you take part in 1 or more companion studies, you will have study visits for this biomarker research study on the following schedule:

* before you start taking the drug(s) if you join a companion drug study and it has been 2 or more weeks since you had these tests done (note: the amount of blood drawn will be about 2 tablespoons at this visit)
* each time you return for imaging scans during the time that you take part in 1 or more companion drug studies
* after you stop taking part in a companion drug study

If your first treatment after consenting to this biomarker research study is part of a clinical research study that is not a companion study or if you receive standard cancer drug(s), you will have study visits for this biomarker research study on the following schedule:

* before you start taking the drug(s) during your first treatment period at MD Anderson and it has been 2 or more weeks since you had these tests done (note: the amount of blood drawn will be about 2 tablespoons at this visit)
* each time you return for imaging scans during your first treatment period at MD Anderson
* after you first stop taking part in a clinical research study that is not a companion drug study, or until you first stop taking standard cancer drug(s).

Length of Treatment:

The study testing will continue:

* for as long as you are taking part in a companion drug study, or
* until you first stop taking part in a clinical research study that is not a companion drug study, or until you first stop taking standard cancer drug(s), if you do not take part in a companion drug study.

Follow-Up Visit:

If you stop taking part in this study:

* You will fill out the cancer symptom questionnaire.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for biomarker, cytokine, and CTC testing.

Long-Term Follow-Up:

After your follow-up visit, from then on, the research staff will collect information on your health status, the drug(s) you receive, and the status of the disease. This information may be collected at the time of standard clinic visits, by reviewing your medical record and imaging scans, and/or by contacting you by phone, mail, and/or email. If you are called, the call will last about 10 minutes or less.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a histologically or cytologically confirmed colorectal adenocarcinoma with metastatic or unresectable, locally advanced disease documented on diagnostic imaging studies.
2. The patient must have been previously treated with systemic chemotherapy for metastatic or unresectable, locally advanced colorectal cancer, with no limit on the number of prior regimens. Patients who develop recurrent or metastatic disease on or within 6 months of adjuvant therapy are eligible.
3. Age >/=18 years to provide a uniform oncologic phenotype of adult-onset colorectal cancer.
4. ECOG performance status 0-2.
5. The patient has signed informed consent.

Exclusion Criteria:

1) Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated with systemic chemotherapy for metastatic colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1275 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Rate of Successful Biomarker Determination | +/- 7 days
  Descriptive analysis performed to report the frequency of informative biomarkers for each of the companion allocation biomarkers as a proportion of patients enrolled onto the study. The primary analysis will be number of patients where informative biomarker results were determined for all tested biomarkers divided by the total number of patients enrolled on the study. Results reported separately for each of the individual biomarkers. Reasons for non-informative results reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Overman MJ, Morris V, Kee B, Fogelman D, Xiao L, Eng C, Dasari A, Shroff R, Mazard T, Shaw K, Vilar E, Raghav K, Shureiqi I, Liang L, Mills GB, Wolff RA, Hamilton S, Meric-Bernstam F, Abbruzzese J, Morris J, Maru D, Kopetz S. Utility of a molecular prescreening program in advanced colorectal cancer for enrollment on biomarker-selected clinical trials. Ann Oncol. 2016 Jun;27(6):1068-1074. doi: 10.1093/annonc/mdw073. Epub 2016 Feb 18. PMID 27045102
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org